CLINICAL TRIAL: NCT03343249
Title: Adjunctive Smart Phone Based Smoking Cessation Treatment
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Texas Southwestern Medical Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: SCCC-PSO1Z14; STU 012014-012 (Other: UTSouthwestern Medical Center)
Record Dates: First submitted 2017-02-09; First posted 2017-11-17 (Actual); Last update posted 2019-01-15 (Actual); Status verified 2019-01

CONDITIONS: High-Risk Cancer

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Study Visits (Experimental): The Short form of the Rapid Estimate of Adult Literacy in Medicine (REALM) will be administered to ensure that all participants are able to read at > sixth grade level. Expired carbon monoxide (CO) will be measured.
  Assessment: Participants will complete self-report questionnaires; and expired CO, weight, and height will be measured. Participants will be provided with a Samsung Galaxy Light Android smart phone and instructed on how to: 1) use the phone features, 2) complete EMAs, and 3) use the adjunctive Smart-T phone based treatment. Participants will receive 4 random prompts and 1 daily diary prompt during their normal waking hours each day for three consecutive weeks. Random assessments will take approximately 1 min to complete and daily diary assessments will take approximately 5 mins to complete.
  Interventions: Behavioral: Smart Phone Based Smoking Cessation

INTERVENTIONS:
Behavioral: Smart Phone Based Smoking Cessation — The Samsung Galaxy Light Smart phone uses the Android 4.2 operating system. The phone has a 4.0 inch (480x800-pixel resolution) touch screen display, a built in microphone, earphone jack, audio speaker, and a rechargeable battery with 12.5 hours of talk time. The phone has 4G and is Wi-Fi and GPS capable. Participants navigate through the EMA program and enter data simply by touching the screen, similar to a pen-and-paper questionnaire. Thus, computer/typing skills are not required. Participants have the ability to call and receive calls from research staff through the smart phone free of charge. All phones will be equipped with Global Positioning Systems (GPS) capability. The smart phones are also equipped with a Secure Digital card to store data as it is collected.

SUMMARY:
Participants will be recruited for the current study during their initial orientation visit to the Parkland Health and Hospital System, Stop Smoking Class and Clinic every Monday morning. Individuals who are interested and eligible for participation in this study will receive uC (Parkland smoking cessation program), plus a tailored, adaptive, smart phone delivered smoking cessation intervention. Participants will be followed weekly from 1 week pre-quit through 4 weeks post-quit. all participants will be asked to attend 6 weekly visits, 4 of these visits will include a thorough assessment that may be completed either before or after their scheduled Parkland treatment appointments. All participants will receive a smartphone at the 1 week pre-quit visit and they will be asked to carry it with them at all times. Participants will complete eMa assessments 5 times per day (4 random assessments + 1 daily dairy) for three consecutive weeks. Geographic location coordinates will be captured during each eMa assessment to link characteristics of the neighborhood environment (e.g., neighborhood socioeconomic status, proximity to tobacco outlets) with cessation-related outcomes. Participants will be compensated upon the return of the smartphone at visit 4 (2 weeks post-quit). Participants will be asked to attend a follow-up visit 12 weeks after their quit date. At this visit, participants will complete additional questionnaires and their smoking status will be assessed. Expired carbon monoxide and weight will also be measured.

DETAILED DESCRIPTION:
Research Supporting Study Objectives. Tobacco use is the leading cause of preventable death in the U.S. Over 443,000 deaths per year are attributable to smoking, with the leading causes of smoking-attributable death being cancer, cardiovascular diseases, and respiratory disease. Although the prevalence of smoking has declined to 20.6% among U.S. adults, 31.1% of those living in poverty are currently smoking. Numerous studies have shown that low SES and financial strain are associated with a reduced likelihood of smoking cessation. As such, lung cancer incidence is far greater among those with low education and who are living in poverty, relative to their higher SES counterparts. Although individuals of low SES are just as likely to attempt smoking cessation, they are less likely to succeed. As such, smoking cessation interventions for low SES populations have had limited success (e.g., biologically confirmed 7-day point prevalence abstinence rates of 7-13% at 6-month follow-up. Innovative smoking cessation interventions are needed to help reduce the rate of smoking in socioeconomically disadvantaged populations of smokers.

Ecological Momentary Assessment and Smoking Cessation Treatments. To date, most studies that have examined smoking and smoking cessation in socioeconomically disadvantaged smokers have used focus groups or traditional lab/clinic based assessment methodology. In the latter scenario, study participants arrive at a lab or clinic for their baseline visit and are asked to answer questions about their "average" or "recent" (e.g., over the past 2 weeks) mood, level of stress, and smoking urges. Participants return to the lab/clinic for follow-up visits and are asked to report thoughts, feelings, and activities that occurred weeks or even months earlier (e.g., "How stressed were you when you smoked your first cigarette after your quit date?"). This type of assessment methodology may result in biased and/or inaccurate estimates due to recall biases and errors in memory and only offers a gross understanding of how cessation symptoms effect smoking lapses and relapse. A more nuanced picture of these symptoms may offer important insights that may be used to create or improve cessation interventions for socioeconomically disadvantaged smokers, who face unique and substantial challenges in quitting smoking.

Ecological momentary assessment (EMA), in which handheld devices (e.g., smart phones) are used to capture moment to moment experience, is currently the most accurate way to measure phenomena in real time in natural settings. EMAs are often used to assess individuals at multiple time points throughout a day. Thus, momentary changes in key variables can be tracked and potentially used to initiate novel interventions. EMA research may facilitate a better understanding of the mechanisms involved in successful cessation attempts, those affecting smoking lapses, and those implicated in the transition from lapse to relapse. Although multiple studies have identified momentary predictors of smoking relapse to our knowledge, no studies have used a participant's responses to EMAs to automatically prompt tailored smoking cessation interventions. Using smart phones to detect high relapse risk situations and automatically deliver tailored smoking cessation treatments may help socioeconomically disadvantaged smokers quit.

ELIGIBILITY:
Inclusion Criteria:

Participants will be included in the study if they:

1. earn a score greater than or equal to 4 on the Short REALM indicating greater than 6th grade English literacy level,
2. are willing to quit smoking 7 days from their first visit,
3. are greater than or equal to 18 years of age,
4. have an expired CO level greater than or equal to 8 ppm suggestive of current smoking,
5. are currently smoking greater than or equal to 5 cigarettes per day,
6. are willing and able to attend 6 weekly sessions (i.e., week -1, quit day, week +1, week +2, week +3, week +4) and the 12 week follow-up session , and
7. have not previously participated in Project PREVAIL [STU 042011-096] at Parkland Hospital. Please note that the Parkland smoking cessation program (usual care) is currently offered in English only.

Exclusion Criteria:

Participants will be excluded from the study if they:

1. are unwilling to quit smoking 7 days from their first visit,
2. have already quit smoking,
3. earn a score less than 4 on the Short REALM indicating less than or equal to 6th grade literacy level,
4. produce an expired CO level less than 8 ppm,
5. are currently smoking less than 5 cigarettes per day,
6. are unwilling or unable to attend 7 assessment sessions,
7. are less than 18 years of age, and/or
8. have not previously participated in Project PREVAIL [STU 042011-096] at Parkland Hospital. Please note that the Parkland smoking cessation program (usual care) is currently offered in English only.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Actual)
Dates: Start 2014-06; Primary Completion 2018-09 (Actual); Study Completion 2018-09 (Actual)

PRIMARY OUTCOMES:
Smoking abstinence | 12 weeks
  Evidence of abstinence from smoking confirmed by questionnaire.

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer Gonzalez, Principal Investigator — University of Texas Southwestern Medical Center

IPD SHARING:
Plan to Share IPD: No